CLINICAL TRIAL: NCT05470777
Title: Safety and Efficacy of CD22/CD19 CAR T-cells and Autologous HSCT Sandwich Strategy as Consolidation Therapy for B-cell Acute Lymphoblastic Leukemia
Brief Title: CD22/CD19 CAR-T and Auto-HSCT Sandwich Strategy as Consolidation Therapy for B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: National Natural Science Foundation of China(Grant No. 81970138) (Unknown); Jiangsu Province Natural Science Foundation of China (Grant No. BK20210091) (Unknown); Jining Medical University (Other); The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Northern Jiangsu People's Hospital (Other); Affiliated Hospital of Nantong University (Other); Suzhou Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Sheng-Li Xue, MD, Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZCART02
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: CD22/CD19 CAR-T; auto-HSCT
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD22/CD19 CAR T and auto-HSCT sandwich strategy as consolidation therapy for B-ALL (Experimental)
  Interventions: Combination Product: CD22/CD19 CAR T and auto-HSCT "sandwich" strategy

INTERVENTIONS:
Combination Product: CD22/CD19 CAR T and auto-HSCT "sandwich" strategy — The patients received sequential infusion of CD22 and CD19 CAR-T cells (co-stimulatory molecule was 4-1BB and infusion dose was 5*10^6/kg respectively) after standard induction and consolidation chemotherapy. Autologous stem cells mobilization and collection were performed 6-8 weeks after CAR-T infusion. Modified BuCy as conditioning regimen for Auto-HSCT was used 4 weeks after successful stem cell collection. CD22 and CD19 CAR-T cells were re-infused 2 days after Auto-HSCT. Patients were followed up and minimal residual diseases (MRD) was monitored by flow cytometry and second-generation gene sequencing of IgH rearrangement.

SUMMARY:
Chimeric antigen receptor T-cell (CAR-T) therapy has achieved remarkable efficacy in B-cell acute lymphoblastic leukemia (B-ALL). However, relapse after CAR-T has been a major issue. Multi-antigen CAR T and combination with other regimens may reduce the relapse rate. The investigators first conducted CD22/CD19 CAR T-cells and auto-HSCT "sandwich " strategy as consolidation therapy in patients with B-ALL. The main Purpose of this study was to observe the safety and efficacy of this new strategy.

DETAILED DESCRIPTION:
The patients received sequential infusion of CD22 and CD19 CAR-T cells (co-stimulatory molecule was 4-1BB and infusion dose was 5*10^6/kg respectively,CAR-T1) after standard induction and consolidation chemotherapy. Autologous stem cells mobilization and collection were performed 6-8 weeks after CAR-T infusion. Standard BuCy as conditioning regimen for Auto-HSCT was used 4 weeks after successful stem cell collection. CD22 and CD19 CAR-T cells were re-infused 2 days after Auto-HSCT(CAR-T2). Patients were followed up and minimal residual diseases (MRD) was monitored by flow cytometry and second-generation gene sequencing of IgH rearrangement.

ELIGIBILITY:
Inclusion Criteria:

* subjects with a primary diagnosis of B-ALL who have any of the following: (a) no suitable allogeneic HSCT donor. (b) refusal of allogeneic HSCT.
* positive expression of CD19 and CD22 in peripheral blood or bone marrow primary cells detected by flow cytometry.
* cardiac ultrasound left ventricular ejection fraction ≥ 50%; Creatinine ≤ 1.6 mg/dl; alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the normal range and total bilirubin ≤ 2.0 mg/dl; Pulmonary function ≤ grade 1 dyspnea (CTCAE v5.0) with oxygen saturation > 91% without oxygenation.
* subjects aged 15-65 years (including 15 and 65 years), regardless of gender.
* T-cell amplification test pass.
* expected survival > 3 months.

Exclusion Criteria:

* patients with recurrence of only isolated extramedullary lesions.
* combination of other malignant tumors.
* previously treated with anti-CD19 or/and CD22 or/and CD3 therapies.
* immunosuppressants use within 2 weeks prior to signing informed consent or plan to immunosuppressants after signing informed consent.
* uncontrolled active infections.
* HIV infection.
* active hepatitis B or hepatitis C infection.
* history of severe tachyphylaxis to aminoglycoside antibiotics.
* history or presence of clinically relevant Central Nervous System (CNS) pathology, such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2020-01-19 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2039-07-21 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  It is measured from the date of the first CAR-T (CAR-T 1) to the date of death from any cause; subjects not known to have died at last follow-up are censored on the date they were last known to be alive

SECONDARY OUTCOMES:
Leukemia-free survival (LFS) | 2 years
  It is measured from the date of achievement of a remission after CAR-T 1 until the date of relapse from CR, or CRi, or death from any cause; subjects not known to have any of these events are censored on the date they were last examined.
Measurable residual disease (MRD) negative rate and duration | 2 years
  MRD is detected by flow cytometry (FC-MRD) and second-generation gene sequencing of IgH rearrangement (NGS-MRD) after the first CAR-T (CAR-T 1) . FC-MRD negative is defined as MRD<10-4 and NGS-MRD negative is defined as MRD<10-6.
Incidence of adverse events (AEs) | 2 years
  AEs will be assessed according to the Common Terminology Criteria for Adverse Events 5.0 (CTCAE5.0) after the first CAR-T (CAR-T 1) .

OTHER OUTCOMES:
Difference in 2-year LFS between the sandwich strategy treatment and external allo-HSCT control group | 2 years
  2-year LFS and 95%CI will be calculated for the sandwich strategy treatment group and external allo-HSCT control group, Log-rank P value will be provided for group comparison result.
Difference in 2-year OS between the sandwich strategy treatment and external allo-HSCT control group | 2 years
  2-year OS and 95%CI will be calculated for the sandwich strategy treatment group and external allo-HSCT control group, Log-rank P value will be provided for group comparison result.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Baseline characteristics of patients and outcome data.
Supporting Information: SAP, CSR
Time Frame: One year after the finishment of the study
Access Criteria: Clinical researchers around the world are all able to access the IPD and supporting information after achieving the authorization of the sponsor. They could be able to get IPD details by visiting ResMan system.
URL: http://www.medresman.org.cn/login.aspx

REFERENCES:
- [Derived] Qian CS, Wang ZH, Li Z, Yao Z, Gong WJ, Wu YJ, Zhou HX, Xu MZ, Qiu Y, Xu SZ, Tan KW, Liu FT, Huang SM, Cao HY, Dai HP, Wu DP, Xue SL. A phase 2 trial of a "sandwich" strategy: Sequential CD22/CD19 chimeric antigen receptor T-cells therapy combined with autologous hematopoietic stem cell transplantation in patients with Philadelphia chromosome-negative B-cell acute lymphoblastic leukemia. Cancer. 2025 Nov 15;131(22):e70168. doi: 10.1002/cncr.70168. PMID 41199560